CLINICAL TRIAL: NCT06953726
Title: CSP #2037T - Veterans Affairs Learning Health System Initiative to Assess Novel Screening vs. Usual Care and Treatment With Apixaban vs. Rivaroxaban in Veterans With Atrial Fibrillation (VALIANT-AF-T) Trial
Brief Title: Comparing the Safety and Efficacy of Apixaban and Rivaroxaban
Acronym: VALIANT-AF-T
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: U.S. Food and Drug Administration (FDA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2037T; 2037 (Other Grant/Funding Number: Veterans Affairs Cooperative Studies Program)
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Ischemic Stroke; Bleeding; Major bleeding
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Hemorrhage | interventions — apixaban; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to twice daily oral administration of apixaban 5mg or daily oral administration of rivaroxaban 20mg. Reduced dose apixaban (2.5 mg twice daily) will be given to participants who meet 2 of the 3 criteria: age 80 years, body weight 60 kg, and serum creatinine 1.5 mg/dL. Reduced dose rivaroxaban (15 mg once daily) will be given to participants with a creatinine clearance 15-50 mL/min.
Masking Description: Drug assignment will be unblinded and distributed through VA's usual mechanism for filling medications (i.e., local pharmacy or Consolidated Mail Outpatient Pharmacy [CMOP]). Randomization will occur via an online tool developed for the study. Each participating site will have a separate block randomization scheme with random block size, programmed into the randomization tool before the start of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apixaban Arm (Active Comparator): Study participants will be randomized to twice daily oral administration of apixaban 5mg. Reduced dose apixaban (2.5 mg twice daily) will be given to participants who meet 2 of the 3 criteria: age 80 years, body weight 60 kg, and serum creatinine 1.5 mg/dL.
  Interventions: Drug: Apixaban
- Rivaroxaban Arm (Active Comparator): Study participants will be randomized to daily oral administration of rivaroxaban 20mg. Reduced dose rivaroxaban (15 mg once daily) will be given to participants with a creatinine clearance 15-50 mL/min.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Apixaban — Study participants will be randomized to twice daily oral administration of apixaban 5mg. Reduced dose apixaban (2.5 mg twice daily) will be given to participants who meet 2 of the 3 criteria: age 80 years, body weight 60 kg, and serum creatinine 1.5 mg/dL.
  Arms: Apixaban Arm
Drug: Rivaroxaban — Study participants will be randomized to daily oral administration of rivaroxaban 20mg. Reduced dose rivaroxaban (15 mg once daily) will be given to participants with a creatinine clearance 15-50 mL/min.
  Arms: Rivaroxaban Arm

SUMMARY:
* The trial will compare two anticoagulants ("blood thinners") that are currently used in the VA and are considered standard care to prevent strokes in patients with atrial fibrillation. The two most commonly-used anticoagulants will be compared: apixaban (Eliquis) and rivaroxaban (Xarelto). They are considered by many doctors to have similar benefits and risks, but no one knows for sure.
* The trial only enrolls patients with a diagnosis of atrial fibrillation ("A Fib").
* The investigators will measure, in about 10,000 VA patients nationally, whether the rates of stroke, major bleeding, or death differ between these two drugs.
* The trial will last about 7 years, but after the first prescription, all information will be collected from electronic medical records.

DETAILED DESCRIPTION:
The study hypothesis is that apixaban will be superior to rivaroxaban with respect to safety using the International Society of Thrombosis and Haemostasis (ISTH) definition of major bleeding and at least non-inferior with respect to efficacy among patients with atrial fibrillation (AF) or atrial flutter (AFL), henceforth noted collectively as "AF". This pragmatic, point-of-care trial will enroll approximately 10,000 Veterans >=age 65 years with AF and a CHA2DS2-VASc score >=3 and randomize them to receive apixaban or rivaroxaban in a 1:1 allocation.

Co-Primary Objectives: Determine in VA trial participants >=age 65 years with non-valvular AF whether oral anticoagulation with apixaban is:

1. Superior to rivaroxaban for the composite safety outcome of ISTH major bleeding
2. Non-inferior to rivaroxaban for the composite efficacy outcome of ischemic stroke, systemic embolism, or all-cause death

Secondary Objectives:

1. Determine in VA trial participants with non-valvular AF whether oral anticoagulation with apixaban is superior to rivaroxaban for the composite efficacy outcome of ischemic stroke, systemic embolism, or all-cause death.
2. Assess impact of anticoagulant therapy on hospitalization for: heart failure, myocardial infarction, or acute coronary syndromes/unstable angina.
3. Examine each component of the composite efficacy endpoint individually (ischemic stroke, systemic embolism, all-cause mortality).

Co-Primary Endpoints:

1. Time to first ISTH-defined major bleeding (Superiority Hypothesis)
2. Time to first ischemic stroke, systemic embolism, or all-cause mortality (Non-Inferiority Hypothesis)

Secondary Endpoints (hierarchically ranked):

1. Time to first ischemic stroke, systemic embolism, or all-cause mortality (Superiority Hypothesis)
2. Time to first ischemic stroke
3. Time to first hospitalization for heart failure, myocardial infarction, or acute coronary syndrome
4. Time to first systemic embolism
5. Time to all-cause death

The estimated number of enrollees will be 10,000 Veterans from approximately 100 VA Medical Centers throughout the U.S.; broad geographical representation in every region is anticipated. Efforts will be made to recruit female Veterans as well as Veterans from diverse racial and ethnic backgrounds with representation of both academic tertiary urban centers and rural community-based outpatient clinics (CBOCs). Strong consideration will be given to selecting enrolling sites based on their prior experience with ambulatory cardiac monitors and, in particular, the 14-day patch monitor (Ziopatch XT), since sites must participate in both the Screening and Treatment Trials. The study will not include enrolling sites outside the U.S.

The primary analysis will comprise Veterans >=65 years, with AF or atrial flutter and CHA2DS2-VASc score >=3. Patients already taking OACs (warfarin or any DOAC) for AF will be eligible. Those on single or dual antiplatelet agents will also be eligible.

Study participants will be randomized to twice daily oral administration of apixaban 5mg or daily oral administration of rivaroxaban 20mg. Reduced dose apixaban (2.5 mg twice daily) will be given to participants who meet 2 of the 3 criteria: age 80 years, body weight 60 kg, and serum creatinine 1.5 mg/dL. Reduced dose rivaroxaban (15 mg once daily) will be given to participants with a creatinine clearance 15-50 mL/min.

The study is planned for 3 years of active enrollment and at least 3 years of remote follow-up of the last enrolled participant, thus 6 years of data collection, with an additional year to completion of data analysis: 7 years (84 months) total.

Enrollment and initiation of anticoagulant will take less than one month for most patients, and up to 90 days for patients randomized to switch to a different OAC who recently received a 90-day supply of their current medication. After randomization to either apixaban or rivaroxaban, all clinical management is per the participants' providers, and all electronic data are collected remotely.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female Veteran, aged 22 years or older
2. Diagnosis of AF or AFL
3. CHADS2VASc >=3
4. Ability to take oral medication and self-reported willingness to adhere to the prespecified apixaban or rivaroxaban regimen

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study; notably use of antiplatelet agents or prior OAC use will not be an exclusion criterion:

1. Current use of oral or injectable anticoagulation, without ability to switch to the assigned study medication
2. Another indication for anticoagulation, such as pulmonary embolism
3. Contraindication to oral anticoagulation
4. Known bleeding diathesis
5. Pregnancy or lactation
6. Known allergic reactions or intolerance to apixaban or rivaroxaban
7. Estimated glomerular filtration rate (eGFR) of < 30 mL/minute
8. Mechanical heart valve
9. Moderate-severe mitral stenosis
10. History of left atrial occlusion, excision, or ligation
11. Current or planned use of ritonavir, itraconazole, or ketoconazole
12. Cardiac or thoracic surgery in the past 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2032-10-04 (Estimated); Study Completion 2033-10-03 (Estimated)

PRIMARY OUTCOMES:
Onset of ISTH Major Bleeding Event | 3 years
  Hospitalization for first ISTH-defined major bleeding, as determined by ICD-10 codes associated with hospitalization. This is the primary safety outcome.
Time to First Stroke | 3 years
  Hospitalization for first stroke, as determined by ICD-10 codes associated with hospitalization. The primary efficacy outcome is time to first event of stroke or systemic embolism, or death of any cause, in days.
Time to First Systemic Embolism | 3 years
  Hospitalization for first systemic embolism, as determined by ICD-10 codes associated with hospitalization. The primary efficacy outcome is time to first event of stroke or systemic embolism, or death of any cause, in days.
Time to All-Cause Mortality | 3 years
  Time to all-cause mortality, as determined by VA data on vital status. The primary efficacy outcome is time to first event of stroke or systemic embolism, or death of any cause, in days.

SECONDARY OUTCOMES:
Time to First Stroke, Systemic Embolism, or All-Cause Mortality | 3 years
  Time to first stroke, systemic embolism, or all-cause mortality (Superiority Hypothesis), as determined by ICD-10 codes associated with hospitalization, or by VA data on vital status.
Time to First Stroke | 3 years
  Time to first stroke, as determined by ICD-10 codes associated with hospitalization. Not part of the Superiority Hypothesis but part of the hierarchically ranked secondary outcome measures.
Time to First Hospitalization for Heart Failure, Myocardial Infarction, or Acute Coronary Syndrome | 3 years
  Time to first hospitalization for heart failure, myocardial infarction, or acute coronary syndrome, as determined by ICD-10 codes associated with hospitalization.
Time to First systemic embolism | 3 years
  Time to first systemic embolism, as determined by ICD-10 codes associated with hospitalization.
All-Cause Mortality | 3 years
  Time to all-cause death, as determined by VA data on vital status.

CONTACTS AND LOCATIONS:
Overall Officials: William E. Boden, MD, Study Chair — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA; Cara N Pellegrini, Study Chair — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No